CLINICAL TRIAL: NCT02257216
Title: A Randomized, Sequential Parallel, Double-Blind, Placebo- Controlled Medical Food Study for the Safety and Efficacy of Vayarin® in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Vayarin® Medical Food Study for Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Vayarin®_006
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2017-01

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1: Treatment/Treatment (Active Comparator): Treatment/Treatment- consists of Vayarin® for 8 weeks followed by 8 weeks of additional treatment with Vayarin®
  Interventions: Other: Vayarin®
- Sequence 2: Placebo/Treatment (Active Comparator): Placebo/Treatment- consists of Placebo for 8 weeks followed by 8 weeks of treatment with Vayarin®
  Interventions: Other: Vayarin®; Other: Placebo
- Sequence 3: Placebo/Placebo (Placebo Comparator): Placebo/Placebo- consists of Placebo for 8 weeks followed by 8 weeks of additional treatment with Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vayarin® — Medical Food
  Arms: Sequence 1: Treatment/Treatment; Sequence 2: Placebo/Treatment
Other: Placebo — Cellulose
  Arms: Sequence 2: Placebo/Treatment; Sequence 3: Placebo/Placebo

SUMMARY:
The primary study objective is to evaluate the efficacy of Vayarin in ADHD adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female age 18-60 inclusive.
2. Primary diagnosis of ADHD
3. At least 50% of the sample will have an abnormal score on the Emotional Control subscale of the BRIEF-A of ≥65.
4. AISRS total score ≥ 24
5. CGI-S ≥4 (moderately ill or worse).
6. Subjects in ongoing psychotherapy will be allowed, but no significant changes in the frequency, type or intensity of the therapy are to be made during the course of their study participation per the discretion of the principal investigator. The subject must be in psychotherapy at least 4 weeks prior to the screening visit.
7. Understands and is able, willing, and likely to fully comply with the study procedures and restrictions.
8. Has given written informed consent to participate in the study.

Exclusion Criteria:

1. BMI less than18.5 or greater than 35.
2. Any underlying/ history or current diagnosis of systemic and/or metabolic disease (e.g. diabetes, Crohn's disease) and/or neurological condition state that may render the subject illegible to participate in the study as assessed by medical history, physical exam, clinical and lab evaluation.
3. History of uncontrolled hypertension or a resting systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg (Subjects with well controlled hypertension on a stable dose (2 months) of anti-hypertensives will be allowed to participate).
4. Hamilton Anxiety Scale (HAM-A) ≥ 17).
5. Hamilton Depression scale (HAM-D ≥ 13).
6. Major depression or anxiety disorder which is a focus of treatment or requires taking medication.
7. A lifetime history of psychosis or bipolar disorder based on a clinician-administered interview using the Mini International Neuropsychiatric Interview (M.I.N.I 7.0). Subjects with mild to moderate forms of social phobia and dysthymia, not requiring treatment, will be allowed.
8. Has any concurrent chronic or unstable medical condition that could confound with the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol.
9. Subjects taking any medication with CNS effects (excluding subjects who discontinue the medications at least 2 weeks prior to the study for stimulants and 4 weeks for SSRI, non-stimulants, and alpha 2-agonist).
10. Subjects with a history of two or more prior failed adequate trials of ADHD treatment due to adverse events.
11. Use of dietary supplements with potential CNS effect, including omega-3 supplements, 30 days before study initiation and throughout the study.
12. Clinical history of cognitive impairment in judgment of investigator.
13. Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed at screening visit prior to randomization. Women of childbearing potential must agree to use adequate birth control for the entire duration of the study.
14. Subjects with a current (within the last 3 months) DSM-V diagnosis of alcohol or drug abuse or dependence (excluding nicotine).
15. Known history of allergic reactions or sensitivity to marine products (fish and seafood), or soy.
16. Has taken an investigational drug or taken part in a clinical trial within 30 days prior to screening.
17. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Adult ADHD Investigator Symptom Rating Scale (AISRS) total score | over 16 weeks

SECONDARY OUTCOMES:
AISRS | over 16 weeks
Adult ADHD Self-Report Scale (ASRS) | over 16 weeks
Clinician Global Impression-Severity (CGI-S) | over 16 weeks
Clinician Global Impression improvement (CGI-I) | over 16 weeks
Behavior Rating Inventory of Executive Function for adults (BRIEF-A) | over 16 weeks
Pittsburgh Sleep Quality Index (PSQI) | over 16 weeks
Adult ADHD Quality of Life Measure (AAQoL) | over 16 weeks
Adverse events monitoring | over 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lenard A Adler, M.D, Principal Investigator — NYU Langone Health; Michael Banov, M.D, Principal Investigator — Northwest Behavioral Research Center; Michael R Liebowitz, M.D, Principal Investigator — The Medical Research Network, LLC; David S Krakow, M.D, Principal Investigator — Bioscience Research, LLC
Locations (4):
- United States (4):
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Bioscience Research, LLC, Mount Kisco, New York
  - New York University School of Medicine, New York, New York
  - The Medical Research Network, LLC, New York, New York